CLINICAL TRIAL: NCT01791595
Title: A Cancer Research UK Phase I Trial of AZD3965, a Monocarboxylate Transporter 1 Inhibitor (MCT1) in Patients With Advanced Cancer
Brief Title: A Phase I Trial of AZD3965 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/12/004; 2010-024463-41 (EudraCT Number)
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Results first posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-02

CONDITIONS: Adult Solid Tumor; Diffuse Large B Cell Lymphoma; Burkitt Lymphoma
Keywords: Phase I; Cancer; Solid Tumours; Diffuse Large B Cell Lymphoma; Monocarboxylate Transporter 1 Inhibitor; lactate; Burkitt Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Neoplasms | interventions — AZD3965

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- AZD3965 Cohort 1 (5 mg OD) (Experimental)
  Interventions: Drug: AZD3965
- AZD3965 Cohort 2 (10 mg OD) (Experimental)
  Interventions: Drug: AZD3965
- AZD3965 Cohort 3 (20 mg OD) (Experimental)
  Interventions: Drug: AZD3965
- AZD3965 Cohort 4 (30 mg OD) (Experimental)
  Interventions: Drug: AZD3965
- AZD3965 Cohort 5 (15 mg BD) (Experimental)
  Interventions: Drug: AZD3965
- AZD3965 Cohort 6 (10 mg BD) (Experimental)
  Interventions: Drug: AZD3965
- AZD3965 Expansion Cohort (10 mg BD) (Experimental)
  Interventions: Drug: AZD3965

INTERVENTIONS:
Drug: AZD3965 — Day -7: single dose of 5 mg AZD3965 orally prior to start of continuous treatment.
  Cycle 1, Day 1: commenced dosing of 5 mg AZD3965 OD orally for up to 6 28-day cycles.
  Trial participants benefitting from treatment could continue beyond 6 cycles for as long as they continued to benefit on agreement between the Investigator and the Sponsor.
  Arms: AZD3965 Cohort 1 (5 mg OD)
Drug: AZD3965 — Day -7: single dose of 10 mg AZD3965 orally prior to start of continuous treatment.
  Cycle 1, Day 1: commenced dosing of 10 mg AZD3965 OD orally for up to 6 28-day cycles.
  Trial participants benefitting from treatment could continue beyond 6 cycles for as long as they continued to benefit on agreement between the Investigator and the Sponsor.
  Arms: AZD3965 Cohort 2 (10 mg OD)
Drug: AZD3965 — Day -7: single dose of 20 mg AZD3965 orally prior to start of continuous treatment.
  Cycle 1, Day 1: commenced dosing of 20 mg AZD3965 OD orally for up to 6 28-day cycles.
  Trial participants benefitting from treatment could continue beyond 6 cycles for as long as they continued to benefit on agreement between the Investigator and the Sponsor.
  Arms: AZD3965 Cohort 3 (20 mg OD)
Drug: AZD3965 — Day -7: single dose of 30 mg AZD3965 orally prior to start of continuous treatment.
  Cycle 1, Day 1: commenced dosing of 30 mg AZD3965 OD orally for up to 6 28-day cycles.
  Trial participants benefitting from treatment could continue beyond 6 cycles for as long as they continued to benefit on agreement between the Investigator and the Sponsor.
  Arms: AZD3965 Cohort 4 (30 mg OD)
Drug: AZD3965 — Day -7: single dose of 30 mg AZD3965 orally prior to start of continuous treatment.
  Cycle 1, Day 1: commenced dosing of 15 mg AZD3965 BD orally for up to 6 28-day cycles.
  Trial participants benefitting from treatment could continue beyond 6 cycles for as long as they continued to benefit on agreement between the Investigator and the Sponsor.
  Arms: AZD3965 Cohort 5 (15 mg BD)
Drug: AZD3965 — Day -7: single dose of 20 mg AZD3965 orally prior to start of continuous treatment.
  Cycle 1, Day 1: commenced dosing of 10 mg AZD3965 BD orally for up to 6 28-day cycles.
  Trial participants benefitting from treatment could continue beyond 6 cycles for as long as they continued to benefit on agreement between the Investigator and the Sponsor.
  Arms: AZD3965 Cohort 6 (10 mg BD)
Drug: AZD3965 — Day -7: single dose of 20 mg AZD3965 orally prior to start of continuous treatment (first 3 trial participants in the Expansion Cohort only; subsequent patients started treatment at Cycle 1, Day 1).
  Cycle 1, Day 1: commenced dosing of 10 mg AZD3965 BD orally for up to 6 28-day cycles.
  Trial participants benefitting from treatment could continue beyond 6 cycles for as long as they continued to benefit on agreement between the Investigator and the Sponsor.
  Arms: AZD3965 Expansion Cohort (10 mg BD)

SUMMARY:
The main aims of this clinical study are to find out the maximum dose that can be given safely to patients, the potential side effects of the drug and how they can be managed and what happens to AZD3965 inside the body.

AZD3965 is a type of drug called a monocarboxylate transporter 1 inhibitor which is being used to stop the growth of cancer cells and kill cancer cells by blocking the action of one of the proteins involved in moving chemical compounds in and out of the cells of the body. This will be the first time that this type of drug has been given to patients.

The drug is a capsule and is taken daily. The study is in two parts. In Part 1 of the study, small groups of patients are treated at increasing doses to find the highest safe dose and best dose to give to patients in Part 2 of the study. It is planned that 40 patients will be entered into Part 1 of the trial.

In Part 2, the dose found to be safe in Part 1 is given to patients with diffuse large B-cell lymphoma (DLBCL) and Burkitt's lymphoma (BL). It is planned that 20 patients will be entered into Part 2 of the trial.

Patients will need to visit the hospital weekly for two months and then every fortnight. Patients will have regular blood and urine tests, scans, heart traces and eye tests amongst other clinical tests. Research blood samples will also be taken to look at what happens to the drug inside the body. Treatment is planned to be given for up to 6 months, but patients benefiting from treatment will be able to keep having it for as long as they continue to benefit. It is important to explain that this is the first study of this drug and patients will have advanced cancer so it is unlikely that patients will benefit directly from taking part but the study may help improve future treatment of cancer.

DETAILED DESCRIPTION:
Part 1 follows a rolling six dose escalation schedule of AZD3965 given once daily (OD) or twice daily (BD) until the maximum tolerated dose (MTD) is defined.

The recommended Phase II dose (RP2D) is based on the safety and pharmacokinetic (PK) results from Part 1.

All patients in Part 2 are treated at this RP2D to further explore the tolerability of this dose and schedule and to explore proof of principle of MCT1 inhibition in tumour types that were shown to express MCT1 and in which AZD3965 showed some effect pre-clinically (DLBCL and BL).

ELIGIBILITY:
Inclusion Criteria:

1. Part 1:

   * Histologically or cytologically proven advanced solid tumour or lymphoma, refractory to conventional treatment or for which no conventional therapy exists.
   * Available archived tumour samples.

   Part 2:
   * Histologically proven DLBCL or BL, which is relapsed or refractory to conventional treatment or for which no conventional therapy exists or has been refused by the patient.
   * Confirmed available tumour samples which can be obtained and used for the study to confirm MCT1 and MCT4 expression as demonstrated by immunohistochemistry.
   * Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or International Working Group (IWG) criteria for Lymphoma.
2. Life expectancy of at least 12 weeks.
3. World Health Organization (WHO) performance status of 0 or 1.
4. Haematological and biochemical indices within the ranges shown below.

   Laboratory Test Value required:
   * Haemoglobin (Hb) ≥9.0 g/dL (90 g/L) or ≥10.0 g/dL (100 g/L) if transfusion within last 4 weeks.
   * Absolute neutrophil count (ANC) Part 1: ≥1.5 x 10^9/L; Part 2: ≥1.0 x 10^9/L.
   * Platelet count Part 1: ≥100 x 10^9/L; Part 2: ≥50 x 10^9/L.
   * Serum bilirubin ≤1.5 x upper limit of normal (ULN).
   * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤2.5 x ULN or ≤5 x ULN in presence of liver metastases (ALP ≤5 x ULN in presence of bone metastases).
   * Glomerular filtration rate (GFR) either: Calculated creatinine clearance or: Isotope clearance measurement (uncorrected) ≥50 mL/min.
   * Prothrombin time <1.5 x ULN.
   * Glucose (fasting) <7.8 mmol/L;
   * Lactate between 0.5 and 2.5 mmol/L inclusive and bicarbonate between 22 mmol/L and 1.5 x ULN inclusive.
5. Left ventricular ejection fraction (LVEF) >50%.
6. 18 years or over.
7. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up.

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C and 4 weeks for investigational medicinal products) before treatment.
2. Ongoing toxic manifestations of previous treatments greater than National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 1. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the Cancer Research UK Centre for Drug Development should not exclude the patient.
3. Symptomatic brain or leptomeningeal metastases.
4. Patients with known retinal disease or macular degeneration affecting visual acuity as assessed by ophthalmologic tests.
5. Female patients who are able to become pregnant (or are already pregnant or lactating). However, those patients who have a negative serum or urine pregnancy test before enrolment and agree to use two forms of contraception (one highly effective form plus a barrier method) [oral, injected or implanted hormonal contraception and condom; intra-uterine device and condom; diaphragm with spermicidal gel and condom] or agree to sexual abstinence, effective from the first administration of AZD3965, throughout the trial and for six months afterwards are considered eligible.
6. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using a barrier method of contraception [condom plus spermicide] or to sexual abstinence effective from the first administration of AZD3965, throughout the trial and for six months afterwards. Men with partners of child-bearing potential must also be willing to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intrauterine device, diaphragm with spermicidal gel or sexual abstinence). Men with pregnant or lactating partners must be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure of the foetus or neonate.
7. Any major surgery in the preceding eight weeks prior to the start of treatment or major thoracic or abdominal surgery from which the patient has not yet recovered.
8. Patients who are unable to swallow oral medication.
9. Alterations to corticosteroid dose within 2 weeks prior to first dose of AZD3965.
10. Gastrointestinal disorders likely to interfere with absorption of the study drug (e.g. partial bowel obstruction or malabsorption).
11. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
12. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV). (N.B. Mandatory testing not required).
13. History of serious allergy or auto-immune disease.
14. Diabetes mellitus (patients with diet controlled diabetes may be included with fasting glucose <7.8 mmol/l and normal haemoglobin A1c [HbA1c]).
15. Cardiac conditions as follows:

    * Clinically significant cardiovascular event within 6 months prior to study entry to include:

      1. acute coronary syndrome (myocardial infarction or unstable angina),
      2. congestive heart failure requiring therapy.
    * Severe valvular heart disease (as defined by British Society of Echocardiography).
    * Presence of an atrial or ventricular arrhythmia, other than atrial fibrillation with well controlled ventricular rate, for which treatment is indicated (anti-arrhythmic drugs or implantable cardioverter defibrillator).
    * Second degree Mobitz type 1 (Wenckebach) heart block with symptoms, or second degree Mobitz type 2 or third degree heart block with or without symptoms unless functioning pacing system.
    * QTc >450 msec in adult male and >460 msec in adult females (QTc to be verified manually [Fridericia's Correction]).
    * History of congenital long QT syndrome.
    * History of Torsade de Pointes (or any concurrent medication with a known risk of inducing QT prolongation).
    * Uncontrolled hypertension (blood pressure ≥160/100 mmHg despite medical therapy).
16. Extensive radiotherapy to greater than 25% of bone marrow within 8 weeks. Prior autologous bone transplant will not exclude a patient.
17. Is a participant, or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study of AZD3965. Participation in an observational or interventional clinical trial that does not involve administration of an IMP would be acceptable.
18. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
19. For Part 2 only: Current malignancies of other types, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri; basal or squamous cell carcinoma of the skin; and patients with low risk prostate cancer on surveillance (with a Gleason score of ≤6 and a Prostate Specific Antigen of ≤10).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Plummer, Prof, Principal Investigator — Freeman Hospital, Newcastle
Locations (7):
- United Kingdom (7):
  - Royal Marsden Hospital, Sutton, London
  - The Beatson West of Scotland, Glasgow, Glasgow
  - Leicester Royal Infirmary, Leicester
  - University College London Hospitals, London
  - The Christie, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noble RA, Bell N, Blair H, Sikka A, Thomas H, Phillips N, Nakjang S, Miwa S, Crossland R, Rand V, Televantou D, Long A, Keun HC, Bacon CM, Bomken S, Critchlow SE, Wedge SR. Inhibition of monocarboxyate transporter 1 by AZD3965 as a novel therapeutic approach for diffuse large B-cell lymphoma and Burkitt lymphoma. Haematologica. 2017 Jul;102(7):1247-1257. doi: 10.3324/haematol.2016.163030. Epub 2017 Apr 6. PMID 28385782
- [Derived] McNeillis R, Greystoke A, Walton J, Bacon C, Keun H, Siskos A, Petrides G, Leech N, Jenkinson F, Bowron A, Halford S, Plummer R. A case of malignant hyperlactaemic acidosis appearing upon treatment with the mono-carboxylase transporter 1 inhibitor AZD3965. Br J Cancer. 2020 Apr;122(8):1141-1145. doi: 10.1038/s41416-020-0727-8. Epub 2020 Feb 20. PMID 32076124
- [Derived] Kershaw S, Cummings J, Morris K, Tugwood J, Dive C. Optimisation of immunofluorescence methods to determine MCT1 and MCT4 expression in circulating tumour cells. BMC Cancer. 2015 May 10;15:387. doi: 10.1186/s12885-015-1382-y. PMID 25957999
- [Derived] Lamb R, Harrison H, Hulit J, Smith DL, Lisanti MP, Sotgia F. Mitochondria as new therapeutic targets for eradicating cancer stem cells: Quantitative proteomics and functional validation via MCT1/2 inhibition. Oncotarget. 2014 Nov 30;5(22):11029-37. doi: 10.18632/oncotarget.2789. PMID 25415228
- See also: Simple summary of trial on Cancer Research UK Trial Database — http://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-trial-azd3965-for-advanced-cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial participants were enrolled at seven trial sites between 23 April 2013 and 24 July 2019. Two additional patients were recruited to the trial but were withdrawn prior to receiving AZD3965.
Period: Part 1 AZD3965 Cohort 1 (5 mg OD)
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
Started | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Evidence of disease progression | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 AZD3965 Cohort 2 (10 mg OD)
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
Started | 0 | 5 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Evidence of disease progression | 0 | 5 | 0 | 0 | 0 | 0 | 0
Period: Part 1 AZD3965 Cohort 3 (20 mg OD)
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
Started | 0 | 0 | 8 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 8 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Evidence of disease progression | 0 | 0 | 6 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 1 AZD3965 Cohort 4 (30 mg OD)
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
Started | 0 | 0 | 0 | 5 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Evidence of disease progression | 0 | 0 | 0 | 2 | 0 | 0 | 0
Period: Part 1 AZD3965 Cohort 5 (15 mg BD)
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
Started | 0 | 0 | 0 | 0 | 11 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 11 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 4 | 0 | 0
Not completed — Evidence of disease progression | 0 | 0 | 0 | 0 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 1 AZD3965 Cohort 6 (10 mg BD)
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
Started | 0 | 0 | 0 | 0 | 0 | 8 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 8 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 5 | 0
Not completed — Evidence of disease progression | 0 | 0 | 0 | 0 | 0 | 3 | 0
Period: Part 2 AZD3965 Expansion (10 mg BD)
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Evidence of disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD) | Total
Number analyzed (Participants) | 3 | 5 | 8 | 5 | 11 | 8 | 11 | 51
Age, Continuous [Median (Full Range); unit: years] | 62 [18 to 75] | 66 [62 to 76] | 64.5 [26 to 77] | 72 [45 to 79] | 63 [22 to 73] | 63.5 [47 to 75] | 70 [48 to 82] | 65 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 2 | 5 | 1 | 4 | 19
  Male | 2 | 2 | 5 | 3 | 6 | 7 | 7 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3 | 5 | 8 | 5 | 11 | 8 | 11 | 51

OUTCOME MEASURES:

1. Primary Outcome: MTD of AZD3965
Description: MTD was determined by testing increasing AZD3965 doses in Part 1 dose escalation cohorts (Cohorts 1-6) and defined as the total daily dose level below that at which ≥2 out of ≤6 evaluable patients had a dose-limiting toxicity (DLT) during Cycle 1 (including Day -7). DLTs were defined as highly probably/probably AZD3965 related haematological, cardiac, ophthalmic, other Grade 3/4 toxicity, death or drug-related toxicity causing AZD3965 interruption >2 weeks (see protocol for specific criteria)
Time Frame: Day -7 to Day 28
Population: All patients recruited to dose escalation cohorts 1 to 6 who received at least one dose of AZD3965 (n=40)
Measure: Number; unit: mg (twice daily)
Groups:
- Part 1 Dose Escalation (Cohorts 1-6): All eligible participants recruited to dose escalation cohorts 1 to 6 who received at least one dose of AZD3965.
Arm/Group | Part 1 Dose Escalation (Cohorts 1-6)
Number analyzed (Participants) | 40
mg (twice daily) | 10

2. Primary Outcome: Number of Patients Who Experienced DLTs
Description: Number of patients who experienced protocol-defined DLTs (defined according to NCI CTCAE version 4.02). DLTs were defined as highly probably/probably AZD3965 related haematological, cardiac, ophthalmic, other Grade 3/4 toxicity, death or drug-related toxicity causing AZD3965 interruption >2 weeks (see protocol for specific criteria)
Time Frame: Day -7 to Day 28
Population: All recruited patients who received at least one dose of AZD3965 (N=51)
Measure: Count of Participants; unit: Participants
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
Number analyzed (Participants) | 3 | 5 | 8 | 5 | 11 | 8 | 11
Participants | 0 | 0 | 1 | 1 | 3 | 2 | 1

3. Primary Outcome: Number of Patients Who Experienced Serious AEs
Description: A serious adverse event (SAE) is any AE, regardless of dose, causality or expectedness, that results in death, is life-threatening, requires in-patient hospitalisation or prolongs existing in-patient hospitalisation, results in persistent or significant incapacity or disability, is a congenital anomaly or birth defect or is any other medically important event. Any ophthalmic and/or cardiac DLT is considered a medically important event and therefore an SAE in this trial. Specific AE terms are provided in the Adverse Events section
Time Frame: From the date of written informed consent and until 28 days after the last dose of AZD3965; an average (median) of 80 days (range: 36 to 517 days)
Population: All recruited patients who received at least one dose of AZD3965 (N=51)
Measure: Count of Participants; unit: Participants
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
Number analyzed (Participants) | 3 | 5 | 8 | 5 | 11 | 8 | 11
Participants | 1 | 1 | 3 | 2 | 8 | 4 | 8

4. Primary Outcome: Number of Patients Who Experienced Non-Serious AEs
Description: A non-serious AE is any untoward medical occurrence that does not meet the serious criteria described for outcome measure 3 above. Specific AE terms are provided in the Adverse Events section
Time Frame: as for outcome 3
Population: All recruited patients who received at least one dose of AZD3965 (N=51)
Measure: Count of Participants; unit: Participants
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
Number analyzed (Participants) | 3 | 5 | 8 | 5 | 11 | 8 | 11
Participants | 3 | 5 | 7 | 5 | 11 | 7 | 11

5. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) From 0 to 24 Hours Post AZD3965 Dosing
Description: Plasma samples were analysed to determine the concentrations of AZD3965 using a previously developed liquid chromatography tandem mass spectrometry (LC-MS/MS) method. For twice daily dosing, Day -7 data reflect the full daily dose but subsequent timepoints reflect half the daily dose as PK sampling was conducted up to 12 hours following the first of the two daily doses; therefore, AUC is from 0 to 12 hours at those timepoints and is reported as a separate outcome measure.
Time Frame: Part 1 (Cohorts 1-4): Day -7 (pre-dose; 0.25, 0.5, 1, 2, 4, 6, 24, 48 hours post-dose) and Day 1 (pre-dose; 0.25, 0.5, 1, 2, 4, 6, 24 hours post-dose)
Population: Part 1: Eligible patients who received AZD3965 on Day -7 and had a baseline and post-dose sample analysed (N=32; could only be calculated for N=5 in Cohort 6 [N=6 for some PK parameters]); Part 2: Eligible patients who received AZD3965 on Day 1 and had a baseline and post-dose sample analysed (N=11). Only calculated for Day -7 and Day 1 in Part 1 and not calculated for other timepoints due to low number of samples or for Part 2 due to limited number of sampling timepoints.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD)
Number analyzed (Participants) | 3 | 5 | 8 | 5 | 6 | 5
h*ng/mL
  Day -7 | 211.7 (84.9) | 730.8 (311.4) | 1509.3 (384.8) | 2843 (1337.4) | 3984.7 (2339.9) | 1540 (693.6)
  Day 1 | 274 (1) | 999 (126.3) | 2123.5 (589.6) | 3031 (1360.5) | NA (NA) — For twice daily dosing, Day -7 data reflect the full daily dose but subsequent timepoints reflect half the daily dose as PK sampling was conducted up to 12 hours following the first of the two daily doses; therefore, AUC is from 0 to 12 hours at those timepoints and is reported as a separate outcome measure | NA (NA) — For twice daily dosing, Day -7 data reflect the full daily dose but subsequent timepoints reflect half the daily dose as PK sampling was conducted up to 12 hours following the first of the two daily doses; therefore, AUC is from 0 to 12 hours at those timepoints and is reported as a separate outcome measure

6. Secondary Outcome: AUC From 0 to 12 Hours Post AZD3965 Dosing
Description: Plasma samples were analysed to determine the concentrations of AZD3965 using a previously developed LC-MS/MS method. AUC from 0 to 12 hours was applicable to twice daily dosing on Day 1 only. See AUC From 0 to 24 Hours Post AZD3965 Dosing for AUC for other cohorts and timepoints.
Time Frame: Part 1 (Cohorts 5-6): Day 1 (pre-dose; 0.25, 0.5, 1, 2, 4, 6, 12 hours post-dose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD)
Number analyzed (Participants) | 6 | 5
h*ng/mL | 1251.5 (654.2) | 620 (272.2)

7. Secondary Outcome: Maximum Observed Plasma Concentration of AZD3965
Description: Plasma samples were analysed to determine the concentrations of AZD3965 using a previously developed LC-MS/MS method. For twice daily dosing, Day -7 data reflect the full daily dose and other timepoints reflect half the daily dose.
Time Frame: Part 1 (Cohorts 1-6): Day -7 (pre-dose; 0.25, 0.5, 1, 2, 4, 6, 24, 48 hours post-dose), Day 1 & 29 (each pre-dose; 0.25, 0.5, 1, 2, 4, 6, 24 hours post-dose [12 hours post-dose if BD]); Part 2 (Expansion): Day 1 (pre-dose; 4, 6, 12 hours post-dose)
Population: Part 1: Eligible patients who received AZD3965 on Day -7 and had a baseline and post-dose sample analysed (N=33) (Only limited samples were available at Day 29); Part 2: Eligible patients who received AZD3965 on Day 1 and had a baseline and post-dose sample analysed (in Part 2 of the trial, PK data were only collected for Day 1)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
Number analyzed (Participants) | 3 | 5 | 8 | 5 | 6 | 6 | 6
ng/mL
  Day -7: number analyzed (Participants) | 3 | 5 | 8 | 5 | 6 | 6 | 0
  Day -7 | 43.4 (22) | 122 (62.7) | 222.7 (95.1) | 377.6 (80.2) | 483.9 (205.7) | 226 (85.7) |
  Day 1 | 38.4 (9.5) | 135.0 (53.2) | 219.9 (62.1) | 458.4 (237) | 213.6 (122.1) | 106.2 (57.1) | 78.5 (42.3)
  Day 29: number analyzed (Participants) | 1 | 2 | 3 | 1 | 0 | 5 | 0
  Day 29 | 48.6 (NA) — Only one patient had evaluable data at this timepoint | 271.6 (123.3) | 310.1 (180.6) | 239.2 (NA) — Only one patient had evaluable data at this timepoint |  | 132.3 (38.6) |

8. Secondary Outcome: Time to Maximum Observed Concentration of AZD3965
Description: as for outcome 7
Time Frame: Part 1 (Cohorts 1-6): Day -7 (pre-dose; 0.25, 0.5, 1, 2, 4, 6, 24, 48 hours post-dose) and Day 1 (pre-dose, 0.25, 0.5, 1, 2, 4, 6, 24 hours post-dose [12 hours post-dose if BD])
Population: Part 1: Eligible patients who received AZD3965 on Day -7 and had a baseline and post-dose sample analysed (N=33); Part 2: Eligible patients who received AZD3965 on Day 1 and had a baseline and post-dose sample analysed (N=11). Only calculated for Day -7 and Day 1 in Part 1; not calculated for other timepoints due to low number of samples or for Part 2 due to number of sampling time points. One patient in Cohort 6 did not have Day -7 data (N=5).
Measure: Median (Full Range); unit: Hour
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD)
Number analyzed (Participants) | 3 | 5 | 8 | 5 | 6 | 6
Hour
  Day -7: number analyzed (Participants) | 3 | 5 | 8 | 5 | 6 | 5
  Day -7 | 1.1 [1 to 2] | 1.1 [1 to 4.1] | 1 [0.5 to 2] | 1.1 [0.5 to 2.1] | 1.5 [0.9 to 4] | 1.92 [0.95 to 4.02]
  Day 1 | 2 [1 to 4] | 2 [1 to 4.2] | 2.05 [1 to 6.1] | 1.1 [1 to 3.9] | 2 [1 to 4] | 1.075 [0.98 to 6.08]

9. Secondary Outcome: Elimination Half Life for AZD3965
Description: Plasma samples were analysed to determine the concentrations of AZD3965 using a previously developed LC-MS/MS method.
Time Frame: Part 1 (Cohorts 1-6): Day -7 (pre-dose; 0.25, 0.5, 1, 2, 4, 6, 24, 48 hours post-dose and Day 1 pre-dose (168 hours post Day -7 dose)
Population: Part 1: Eligible patients who received AZD3965 on Day -7 and had a baseline and post-dose sample analysed (N=32; one patient had a reduced dose in Cohort 6 at Day -7 so these data are not included in half life calculation). Not calculated for Part 2 due to limited number of sampling timepoints.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD)
Number analyzed (Participants) | 3 | 5 | 8 | 5 | 6 | 5
Hour | 51.9 (4.9) | 45.4 (6.4) | 38.3 (5.9) | 38.7 (13.3) | 37.5 (8.5) | 33.6 (4.3)

10. Secondary Outcome: Plasma Level of Cell Death Marker M30 (Caspase-Cleaved CK18; Part 1 Only)
Description: Plasma samples were analysed to determine the level of M30 using a validated cell death ELISA in Part 1 (Cohorts 1-6). Assays not conducted for Part 2 of the trial as considered uninformative.
Time Frame: Baseline (Day -14 to -8), Day -7 (pre-dose) Day 1 (24 hours post-dose), Day 8 (pre-dose), Day 29 (pre-dose)
Population: All patients in Part 1 who received AZD3965 and provided pre and post-treatment blood samples (N=37). Some patients did not have data at all timepoints
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD)
Number analyzed (Participants) | 3 | 5 | 8 | 5 | 11 | 5
U/L
  Baseline: number analyzed (Participants) | 1 | 4 | 8 | 5 | 11 | 5
  Baseline | 383 (NA) — Only one patient had evaluable data at this timepoint | 944.8 (72.6) | 392.3 (300.3) | 196.0 (96.3) | 464.9 (304.9) | 359.6 (364)
  Day -7: number analyzed (Participants) | 2 | 5 | 8 | 5 | 11 | 5
  Day -7 | 201 (17) | 865.6 (250.3) | 410.1 (296.5) | 225.6 (114.5) | 464.8 (312.3) | 342 (371.9)
  Day 1: number analyzed (Participants) | 2 | 5 | 8 | 5 | 11 | 5
  Day 1 | 174.5 (60.1) | 860.6 (191.5) | 428.4 (302.9) | 220.6 (112.7) | 487.9 (326.9) | 336.6 (375.9)
  Day 8: number analyzed (Participants) | 3 | 5 | 7 | 5 | 9 | 5
  Day 8 | 226 (86.2) | 959.4 (90.8) | 457.1 (339.5) | 206.8 (90.2) | 418.6 (327.8) | 343.4 (370.8)
  Day 29: number analyzed (Participants) | 2 | 3 | 5 | 4 | 3 | 5
  Day 29 | 176 (46.7) | 836.7 (282.9) | 428 (366.6) | 267.8 (157.8) | 660.3 (489.7) | 344.6 (369.5)

11. Secondary Outcome: Plasma Level of Cell Death Marker M65 (Total Plus Caspase-Cleaved CK18; Part 1 Only)
Description: Plasma samples were analysed to determine the level of M65 using a validated cell death enzyme-linked immunosorbent assay (ELISA) in Part 1 (Cohorts 1-6). Assays not conducted for Part 2 of the trial as considered uninformative.
Time Frame: Baseline (Day -14 to -8), Day -7 (pre-dose) Day 1 (24 hours post-dose), Day 8 (pre-dose), Day 29 (pre-dose)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD)
Number analyzed (Participants) | 3 | 5 | 8 | 5 | 11 | 5
U/L
  Baseline: number analyzed (Participants) | 1 | 4 | 8 | 5 | 11 | 5
  Baseline | 533.0 (NA) — Only one patient had evaluable data at this timepoint | 4496.0 (1008.0) | 1602.1 (1627.4) | 1046.6 (1338.7) | 1344.3 (1202.5) | 287.6 (192.2)
  Day -7: number analyzed (Participants) | 2 | 5 | 8 | 5 | 11 | 5
  Day -7 | 623.5 (446.2) | 3846.4 (1772.5) | 1796.4 (1697.6) | 935.6 (1000.7) | 1488.7 (1409.6) | 233.2 (126.9)
  Day 1: number analyzed (Participants) | 2 | 5 | 8 | 5 | 11 | 5
  Day 1 | 469.0 (12.7) | 3935.6 (1522.0) | 1742.0 (1840.9) | 981.0 (1054.8) | 1673.0 (1450.2) | 255.4 (157.3)
  Day 8: number analyzed (Participants) | 3 | 5 | 7 | 5 | 9 | 5
  Day 8 | 841.3 (651.4) | 4478.4 (730.2) | 1807.0 (2072.6) | 474.2 (568.5) | 1418.4 (1472.6) | 252.0 (155.1)
  Day 29: number analyzed (Participants) | 2 | 3 | 5 | 4 | 3 | 5
  Day 29 | 801.5 (314.7) | 5000.0 (0.0) | 1226.8 (2123.2) | 443.0 (566.5) | 2609.3 (2452.2) | 285.0 (172.3)

12. Secondary Outcome: Plasma Level of Nucleosomal DNA (nDNA) as a Measure of Apoptosis (Part 1 Only)
Description: Plasma samples were analysed to determine the level of nDNA using validated methodology in Part 1 (Cohorts 1-6). Assays not conducted for Part 2 of the trial as considered uninformative.
Time Frame: Baseline (Day -14 to -8), Day -7 (pre-dose) Day 1 (24 hours post-dose), Day 8 (pre-dose), Day 29 (pre-dose)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Optical density
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD)
Number analyzed (Participants) | 3 | 5 | 8 | 5 | 11 | 5
Optical density
  Baseline: number analyzed (Participants) | 1 | 4 | 8 | 5 | 11 | 5
  Baseline | 0.123 (NA) — Only one patient had evaluable data at this timepoint | 0.778 (1.144) | 0.614 (0.865) | 0.170 (0.138) | 0.485 (0.879) | 0.139 (0.134)
  Day -7: number analyzed (Participants) | 2 | 5 | 8 | 5 | 11 | 5
  Day -7 | 0.450 (0.180) | 0.731 (0.860) | 0.580 (0.889) | 0.204 (0.187) | 0.259 (0.257) | 0.140 (0.158)
  Day 1: number analyzed (Participants) | 2 | 5 | 8 | 5 | 11 | 5
  Day 1 | 0.397 (0.372) | 0.924 (1.114) | 0.593 (0.796) | 0.200 (0.186) | 0.241 (0.191) | 0.140 (0.146)
  Day 8: number analyzed (Participants) | 3 | 5 | 7 | 5 | 9 | 5
  Day 8 | 0.441 (0.280) | 1.111 (1.059) | 0.697 (1.033) | 0.206 (0.135) | 0.287 (0.305) | 0.149 (0.136)
  Day 29: number analyzed (Participants) | 2 | 3 | 5 | 4 | 3 | 5
  Day 29 | 0.298 (0.270) | 1.060 (0.538) | 0.841 (1.208) | 0.144 (0.116) | 0.195 (0.179) | 0.156 (0.144)

13. Secondary Outcome: Number of Patients Who Experienced a Complete Response, Partial Response or Stable Disease According to RECIST 1.1 or a Complete Remission, Partial Remission or Stable Disease According to the IWG Criteria for Lymphoma (Part 2 Only)
Description: Antitumour activity measured according to RECIST version 1.1 (solid tumours)(see Eishenhauer et al; Eur J Cancer 2009, 45:228-247) or IWG criteria for Lymphoma (lymphoma)(see Cheson, Fisher et al; JCO 2014, 32:3059-3067). Complete or partial response/remission was confirmed by repeat measurements ≥4 weeks after response criteria were met; patients with stable disease met criteria at least once ≥6 weeks after first dose of AZD3965
Time Frame: Radiological disease assessment at screening/baseline and every 6 weeks to end of treatment; an average (median) of 44 days (range: 36 to 432 days)
Population: Part 2: All patients who met the eligibility criteria, received at least 75% of their first continuous treatment cycle (28 days) and had a baseline assessment of disease (N=5)
Measure: Count of Participants; unit: Participants
Arm/Group | AZD3965 Expansion Cohort (10 mg BD)
Number analyzed (Participants) | 5
Participants
  Stable disease | 1
  Complete remission | 1

ADVERSE EVENTS:
Time Frame: Safety data was collected from the date of written informed consent and continued until 28 days after the last dose of AZD3965, an average (median) of 80 days (range: 36-517).
Description: AE terms from vocabulary, NCI CTCAE V4.02 for Part 1 (AZD3965 Cohorts 1-6) and MedDRA V23.0 for Part 2 (Expansion Cohort)
Groups:
- AZD3965 Expansion Cohort (10 mg BD): AZD3965: Day -7: single dose of 20 mg AZD3965 orally prior to start of continuous treatment (first 3 trial participants in the Expansion Cohort only; subsequent patients started treatment at Cycle 1, Day 1).
  Cycle 1, Day 1: commenced dosing of 10 mg AZD3965 BD orally for up to 6 28-day cycles.
  Patients benefitting from treatment could continue beyond 6 cycles for as long as they continued to benefit on agreement between the Investigator and the Sponsor.
Arm/Group | AZD3965 Cohort 1 (5 mg OD) | AZD3965 Cohort 2 (10 mg OD) | AZD3965 Cohort 3 (20 mg OD) | AZD3965 Cohort 4 (30 mg OD) | AZD3965 Cohort 5 (15 mg BD) | AZD3965 Cohort 6 (10 mg BD) | AZD3965 Expansion Cohort (10 mg BD)
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/5 | 0/8 | 0/5 | 0/11 | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/5 | 3/8 | 2/5 | 8/11 | 4/8 | 8/11
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 7/8 | 5/5 | 11/11 | 7/8 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD3965 Cohort 1 (5 mg OD) (N=3) | AZD3965 Cohort 2 (10 mg OD) (N=5) | AZD3965 Cohort 3 (20 mg OD) (N=8) | AZD3965 Cohort 4 (30 mg OD) (N=5) | AZD3965 Cohort 5 (15 mg BD) (N=11) | AZD3965 Cohort 6 (10 mg BD) (N=8) | AZD3965 Expansion Cohort (10 mg BD) (N=11)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD3965 Cohort 1 (5 mg OD) (N=3) | AZD3965 Cohort 2 (10 mg OD) (N=5) | AZD3965 Cohort 3 (20 mg OD) (N=8) | AZD3965 Cohort 4 (30 mg OD) (N=5) | AZD3965 Cohort 5 (15 mg BD) (N=11) | AZD3965 Cohort 6 (10 mg BD) (N=8) | AZD3965 Expansion Cohort (10 mg BD) (N=11)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (3) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 3 (4) | 3 (3) | 2 (6) | 4 (4) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 2 (2) | 2 (2) | 4 (4) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blindness transient (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin T increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (4) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ear pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 5 (5) | 5 (5)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genitals enlarged (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
H3N2 influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 2 (5) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 2 (3) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Moraxella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 1 (1) | 2 (4) | 3 (3) | 1 (1) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 2 (3) | 5 (7) | 4 (6) | 2 (3) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 3 (4) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (4) | 0 (0) | 1 (3) | 4 (4) | 2 (2) | 2 (2)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Lactate accumulation in peripheral blood mononuclear cells was originally a measure for assessment of the primary objective but the assay was confounded by methodological problems and high inter-patient variability. This measure was removed for Part 2 and not used for assessment of the primary objective. M30, M65 and nDNA assays are only quasi quantitative; data >upper limit substituted with upper limit and data <lower limit substituted with lower limit/2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT01791595/Prot_000.pdf